CLINICAL TRIAL: NCT06181240
Title: Modification of Coronary Calcium With Laser Based Intravascular Lithotripsy for Coronary Artery Disease (FRACTURE)
Acronym: FRACTURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolt Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-005614
Record Dates: First submitted 2023-11-22; First posted 2023-12-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Calcification
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, single-arm, multicenter, interventional study in adults (≥18 years of age) with de novo, calcified, stenotic coronary artery lesions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Bolt IVL System (Experimental): Lithotripsy is a medical procedure that uses shock waves to modify intravascular calcium.
  Interventions: Device: Intravascular lithotripsy

INTERVENTIONS:
Device: Intravascular lithotripsy — Lithotripsy-enhanced percutaneous coronary intervention of de novo, calcified, stenotic coronary artery lesions prior to stenting.

SUMMARY:
The FRACTURE Trial is a prospective, non-randomized, single-arm, multicenter, interventional study in US and international centers.

DETAILED DESCRIPTION:
The FRACTURE Trial is a prospective, non-randomized, single-arm, multicenter, interventional study in US and international centers with the Bolt Intravascular Lithotripsy System that was designed to percutaneous transluminal angioplasty by utilizing delivery of IVL to disrupt calcium prior to full balloon dilatation at low pressures.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is ≥18 years of age;
* Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for Percutaneous Coronary Intervention (PCI);
* For patients with unstable ischemic heart disease, a local site-based biomarker (preferably troponin or hs-troponin) must be less than or equal to the upper limit of lab normal (ULN) within 12 hours prior to the study procedure;
* For patients with stable ischemic heart disease, CK-MB will be drawn at the time of the study procedure from the side port of the sheath; results need not be analyzed prior to enrollment, but must be less than or equal to the upper limit of lab normal (ULN);
* Single de novo target lesion stenosis of protected LMCA, or LAD, RCA, or LCX (or of their branches) with:

  * Stenosis of ≥70% and <l00%; or
  * Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.90, or IVUS or OCT minimum lumen area ≤4.0 mm2;
* Evidence of calcification at the target lesion site by

  * angiography, with fluoroscopic radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, or
  * Intravascular Ultrasound (IVUS) or Optical Coherence Tomography (OCT), with presence of ≥270 degrees of calcium on at least 1 cross section;
* Ability to pass a 0.014" guidewire across the lesion.

Key Exclusion Criteria:

* Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure;
* New York Heart Association (NYHA) class III or IV heart failure at time of index procedure;
* Prospective need for hemodynamic support, i.e., IABP or Impella;
* Chronic kidney disease with serum creatinine >2.5 mg/dL, eGFR <30 mL/min/1.73m2, or on chronic dialysis;
* Unprotected left main diameter stenosis >50%;
* Target vessel is excessively tortuous defined as the presence of two or more bends >90º or three or more bends >75º;
* Target lesion is an ostial location (LAD, LCX, or RCA, within 5 mm of ostium) or an unprotected left main lesion;
* Chronic Total Occlusion;
* Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-02-09 (Actual); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Within 30 days following procedure
  Freedom from major adverse cardiac events (MACE) within 30 days following the index procedure.
Primary Effectiveness Endpoint | Immediately after the intervention/procedure/surgery
  Procedural success defined as successful stent delivery with a final residual stenosis <50% (assessed by angiographic core laboratory) and freedom from in-hospital MACE.

SECONDARY OUTCOMES:
Device success | Immediately after the intervention/procedure/surgery
  The ability to deliver the Bolt IVL catheter across the target lesion, and delivery of lithotripsy without serious angiographic complications immediately after IVL.
Angiographic success (at <50%) | Immediately after the intervention/procedure/surgery
  Stent delivery with <50% final residual stenosis and without serious angiographic complications.
Procedural success | Immediately after the intervention/procedure/surgery
  Stent delivery with a final residual stenosis ≤30% and without in-hospital MACE.
Angiographic success (at ≤30%) | Immediately after the intervention/procedure/surgery
  Stent delivery with ≤30% final residual stenosis and without serious angiographic complications.
Serious angiographic complications | Immediately after the intervention/procedure/surgery
  Severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
MACE | within 6, 12, and 24 months.
  MACE within 6, 12, and 24 months.
Target lesion failure (TLF) | 30 days, 6 months, 12 months, and 24 months
  Cardiac death, target vessel myocardial infarction (TV-MI) (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods at 30 days, 6 months, 12 months, and 24 months.
All deaths, cardiac deaths, MIs, TV-MIs, procedural and nonprocedural MIs, ID-TVRs, ID-TLRs, non-ID-TLRs, non-ID-TVRs, all revascularizations (ID and non-ID), and stent thrombosis | Periprocedure, within 30 days, 6 months, 12 months, and 24 months
  All deaths, cardiac deaths, MIs, TV-MIs, procedural and nonprocedural MIs, ID-TVRs, ID-TLRs, non-ID-TLRs, non-ID-TVRs, all revascularizations (ID and non-ID), and stent thrombosis (Academic Research Consortium (ARC) definite, probable, definite or probable).

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McEntegart, MD, PhD, Principal Investigator — NY Presbyterian Hospital/Columbia University Medical Center; Nicholas van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (46):
- United States (31):
  - Scripps Health, La Jolla, California
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Riverside Community Hospital, Riverside, California
  - Southern California Permanente Medical Gp. / Kaiser Permanente, San Diego, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Nova Clinical Research Centers/Manatee Memorial Hospital, Bradenton, Florida
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - HCA FL Memorial Hospital, Jacksonville, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Research Institute, Hiram, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Metropolitan Heart and Vascular Institute, Coon Rapids, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The Valley Hospital, Paramus, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - The Icahn School of Medicine at Mt. Sinai, New York, New York
  - Nyph/Cuimc, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Providence Heart Institute, Portland, Oregon
  - Wellspan York Hospital, York, Pennsylvania
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - Austin Heart Research, Austin, Texas
  - Methodist Healthcare Methodist Research Institute, San Antonio, Texas
  - Intermountain Health, Murray, Utah
  - Chippenham Johnson Willis Hospital, Richmond, Virginia
- Onze-Lieve-Vrouwziekenhuis, afgekort OLV ziekenhuis, Aalst, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- Germany (3):
  - Segeberger Kliniken GmbH,, Bad Segeberg
  - Cellitinnen Krankenhaus St. Vinzenz, Cologne
  - SJG St. Paulus GmbH, St.-Johannes-Hospital Dortmund, Dortmund
- Lithuania (2):
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Netherlands (2):
  - Amsterdam University Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
- United Kingdom (6):
  - Harefield Hospital, Harefield
  - Royal Free Hospital, London
  - St. Thomas' Hospital, London
  - King's College Hospital, London
  - St George's University of London, London
  - Royal Brompton Hospital, London